CLINICAL TRIAL: NCT00723697
Title: Etude Observationnelle Prospective de l'Utilisation en Situation Reelle; Prospective Real Situation Observational Study of Subutex® or Its Buprenorphine High Dose Generic (BHD) in the Replacement Treatment of Major Opiate Dependence: Following Parameters With Respect to Misuse and Pharmacovigilance
Brief Title: Observational Study of Misuse of High Dose Buprenorphine (Subutex® or Generic) in Opiate-Addicted Patients in France (Study P05186AM1)(COMPLETED)
Acronym: OPUS R
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P05186
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Buprenorphine; Naloxone; Opiate-related Disorders; Opiate Dependence; Drug Abuse
Keywords: Subutex
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine; Drugs, Generic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients addicted to opiates and requiring replacement treatment. Patients in this non-interventional study were prescribed treatment as per usual clinical practice.
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — 0.4, 2, or 8 mg sublingual tablets
  Other Names: Subutex; buprenorphine high dose (BHD) generic (Arrow Laboratories); SCH 028444

SUMMARY:
The purpose of this study is to assess the risks of abuse, misuse and adverse events related to high dose buprenorphine. Approximately 1250 patients taking Subutex (Schering-Plough) or its Buprenorphine High Dose (BHD) generic (Arrow Laboratories) will participate in this study. Data will be collected using physician questionnaires and self evaluation patient questionnaires at the first visit and visits at 6 and 12 months.

DETAILED DESCRIPTION:
Approximately 380 physicians will participate in this study. Patients will be enrolled in chronological order of consultations.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be those already having a prescription for Subutex or its BHD generic, or being proposed a prescription for Subutex or its BHD generic for the first time when consulting the participating physician.
* The patient must have been informed orally and in writing via the information notice and have signed it.

Exclusion Criteria:

* Criteria of non-eligibility will be related to the contraindications in the Marketing Authorization (MA) of Subutex or its BHD generic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients addicted to opiates and requiring replacement treatment with Subutex (Schering-Plough) or BHD generic (Arrow laboratories)
Sampling Method: Non-Probability Sample
Enrollment: 1307 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 1307
Completed | 1289
Not Completed | 18
Not completed — Physician questionnaires not received | 2
Not completed — Missing Informed Consent Form | 10
Not completed — Other exclusion criteria applied | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 879
Age, Continuous [Mean (Full Range); unit: years] — A total of 880 patients returned a Day 1 self-questionnaire; only 824 patients had identifiable ages.
  years | 34.70 [14 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — A total of 880 patients returned a Day 1 self-questionnaire; 879 patients had identified gender.
  Participants
    Female | 192
    Male | 687

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Misuse (Injection, Sniffing, Dose Fractionation, Modification of Prescribed Doses, and Combination With Psychotropic Agents)
Description: Number of patients who indicate misuse behaviours on self-questionnaire response at first (D1), 6 month (M6), and 12 month (M12) visits.
Time Frame: first visit, 6 months, and 12 months
Population: Number of patients with self-questionnaire responses.
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 880
participants
  Proper usage at all visits (no misuse) | 131 [30.61 to 39.57]
  Misuse at M12 only | 20
  Misuse at M6 only | 15
  Misuse at D1 only | 38
  Misuse at M6 and M12 only | 19
  Misuse at D1 and M12 only | 24
  Misuse at D1 and M6 only | 34
  Misuse at all visits | 151
  Missing Data | 448

2. Secondary Outcome: Number of Patients Reporting Clinical Consequences of Engaging in Misuse
Description: Number of patients with clinical consequences (development or progression of: abscess, nutritional deficiency, dental problems, psychiatric problems including depression, sleep problems, schizophrenia, anxiety, phobias, hallucinations, delirium, withdrawal symptoms, inhibition, suicide attempts and other problems) at first, 6 month, and/or 12 month visit.
Time Frame: first visit, 6 months, and 12 months
Population: Number of patients analyzed for the consequence, at each visit.
Measure: Number; unit: participants
Groups:
- Patients at First Visit; Patients at 6 Month Visit; Patients at 12 Month Visit: Patients addicted to opiates and requiring replacement treatment. Patients in this non-interventional study were prescribed treatment as per usual clinical practice.
Arm/Group | Patients at First Visit | Patients at 6 Month Visit | Patients at 12 Month Visit
Number analyzed (Participants) | 1289 | 1136 | 1024
participants
  abscesses (n=1288/1134/1022) | 41 | 29 | 31
  nutritional deficiency (n=1288/1134/1022) | 99 | 65 | 63
  dental problems (n=1287/1133/1022) | 459 | 293 | 244
  psychiatric problems (n=1288/1133/1022) | 504 | 364 | 329
  depression (n=502/359/325) | 230 | 174 | 157
  schizophrenia (n=499/356/326) | 18 | 15 | 15
  sleep disturbances (n=500/360/327) | 336 | 228 | 200
  anxiety (n=500/360/326) | 335 | 222 | 200
  delirium/hallucinations (n=499/358/327) | 26 | 21 | 17
  autistic withdrawal, inhibition (n=500/357/326) | 89 | 50 | 43
  suicide attempts (n=499/357/326) | 42 | 14 | 12
  other psychiatric problems (n=487/355/326) | 28 | 14 | 18

3. Primary Outcome: Number of Patients With Misuse (Injection, Sniffing, Dose Fractionation, Modification of Prescribed Doses, and Combination With Psychotropic Agents) as Reported by Physician.
Description: Number of patients with misuse behaviours on physician-questionnaire response at first (D1), 6 month (M6), and 12 month (M12) visits.
Time Frame: first visit, 6 months, and 12 months
Population: All eligible patients
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 1289
participants
  Proper usage at all visits (no misuse) | 206
  Misuse at M12 only | 37
  Misuse at M6 only | 37
  Misuse at D1 only | 134
  Misuse at M6 and M12 only | 52
  Misuse at D1 and M12 only | 49
  Misuse at D1 and M6 only | 72
  Misuse at all visits | 407
  Missing Data | 295

ADVERSE EVENTS:
Description: Two patients who did not have a first visit were excluded from the adverse event database.
Arm/Group | Patients
Serious Adverse Events (participants affected / at risk) | 34/1305
Other Adverse Events (participants affected / at risk) | 0/1305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=1305)
CARDIAC DISORDER (Cardiac disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL STENOSIS (Gastrointestinal disorders) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1)
INJECTION SITE NECROSIS (General disorders) | 5 (8)
OEDEMA (General disorders) | 6 (7)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1)
INJECTION SITE ABSCESS (Infections and infestations) | 9 (10)
PSOAS ABSCESS (Infections and infestations) | 1 (1)
TUBERCULOSIS (Infections and infestations) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (3)
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 (1)
DRUG DEPENDENCE (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
MENTAL DISORDER (Psychiatric disorders) | 7 (7)
WITHDRAWAL SYNDROME (Psychiatric disorders) | 3 (3)
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALCOHOL USE (Social circumstances) | 1 (1)
DRUG DETOXIFICATION (Surgical and medical procedures) | 2 (2)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication (abstract, poster, communication...) can be made without the agreement of SCHERING-PLOUGH.